CLINICAL TRIAL: NCT03506321
Title: Comparative Analysis of the Incremental Benefit of Chromoendoscopy in Addition to High Definition White Light (HD-WL)and Narrow Band Imaging (NBI) for the Prediction of Submucosal Invasive Cancer Within Laterally Spreading Lesions (LSLs) and in Determining the Presence of Residual or Recurrent Adenoma at a Post Endoscopic Resection Scar
Brief Title: Comparison of the Benefit of Chromoendoscopy in Addition to High Definition White Light and Narrow Band Imaging for the Prediction of Submucosal Invasive Cancer in Colonic Lesions
Acronym: LANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HREC/16/WMEAD/392(4863)
Record Dates: First submitted 2018-03-13; First posted 2018-04-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colonic Adenoma; Colon Polyp; Submucosal Invasive Colon Adenocarcinoma; Colorectal Cancer
Keywords: colonoscopy; Residual adenoma; Recurrent adenoma
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms; Adenoma | interventions — Narrow Band Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LANS (Other): Lesions are assessed with chromoendoscopy, HD-WL & NBI
  Interventions: Diagnostic Test: chromoendoscopy, high definition white light and narrow band imaging

INTERVENTIONS:
Diagnostic Test: chromoendoscopy, high definition white light and narrow band imaging — Chromoendoscopy, high definition white light and narrow band imaging are compared for predicting submucosal invasion within laterally spreading lesions in the colon and determining the presence of residual or recurrent adenoma at the post endoscopic resection scar

SUMMARY:
To compare the incremental benefit of chromoendoscopy in addition to high definition white light and narrow band imaging in predicting submucosal invasion within laterally spreading lesions in the colon and in determining the presence of residual or recurrent adenoma at the post endoscopic resection scar

DETAILED DESCRIPTION:
Wide-field (WF) EMR is now accepted as a safe and effective alternative to surgery for removal of large (>20mm) laterally spreading lesions (LSLs).

Assessment of the risk of submucosal invasive cancer (SMIC) is paramount to determining whether a lesion should be attempted for resection by endoscopic mucosal resection (EMR). Lesions that are at high risk for invading the submucosa should either be referred for surgery or in selected cases may be removed by endoscopic submucosal dissection (ESD) in an en bloc fashion to assess SMIC accurately. Tools to assess the likelihood of SMIC endoscopically include analysis of the Kudo pit-pattern (KPP) combined with assessment of morphology as per Paris classification.

KPP analysis is useful to predict histology based on the microarchitecture of pits, epithelial crests or ridges. It thus provides an assessment of risk of sub-mucosal invasion of superficial lesions. There are five categories; with Type 1 and 2 being non-tumours i.e. benign lesion, as compared to Type 3-5 which are tumours ranging from pre-cancerous adenomas (tubular or villous adenoma) to invasive cancer.

Assessment of lesion morphology at WF-EMR using the Paris Classification and analysis of the surface pit-pattern are an integral part of identifying lesions suitable for EMR.

As per the Paris Classification superficial lesions in the colon are divided into; polypoid, non-polypoid and mixed types. Non-polypoid lesions are further divided into slightly raised (0-IIa), flat (0-IIb), depressed surface (0-IIc) or mixed types such as a flat lesion with a nodule (0-IIa+b). The later generally have a greater risk for sub-mucosal invasion (SMI) than polypoid lesions and can be as high as 35-40%. Flat lesions are referred to as laterally spreading lesions (LSLs) if greater than 10mm. There are two distinct subtypes; non-granular vs granular. Granular LSLs exhibit a lower risk of SMI as compared to non-granular LSLs.

Expert opinion suggests that differentiating the KPP in large LSLs (>20mm) requires chromoendoscopy or magnifying endoscopy. This can be a time intensive process. New advances in optics focusing on manipulating the wavelength of the light source; e.g. narrow band imaging (NBI) with the Olympus platform or Fujinon intelligent colour enhancement (FICE) with Fuji have become readily available, and show potential, particularly when combined with magnification, in discriminating the KPP and therefore predicting risk for SMIC. These technologies essentially provide virtual chromoendoscopy. Their diagnostic accuracy has been shown to be comparable to indigo-carmine chromoendoscopy. Both chromoendoscopy and NBI have shown superiority in accurately differentiating between neoplastic and non-neoplastic lesions as compared to high definition white light (HD-WL) endoscopy. In addition NBI has been shown to have a negative predictive value of 98% in assessing residual or recurrent adenoma (RRA) at an EMR scar.

No studies to date have assessed the use of chromoendoscopy and the subsequent benefit of high-definition imaging (HD-WL + NBI) in predicting SMIC and RRA at an EMR scar.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to give informed consent to involvement in trial. For patients who do not speak English, an interpreter will be asked to translate the informed consent
* Patients referred to Westmead and Auburn Hospital Endoscopy Unit for a colonoscopy for all indications

Exclusion Criteria:

* Patient's with known colonic strictures/stenosis
* Patient's with active inflammatory bowel disease
* Pregnancy
* Patients who did not consent to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2021-03-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Compare chromoendoscopy predictions and HD-WL/NBI predictions of submucosal invasive cancer (SMIC) and residual or recurrent adenoma (RRA) to compare correlation with histological findings | Three years

SECONDARY OUTCOMES:
Accurate histologic correlation as predicted by Kudo pit pattern classification | Three years
Compare inter-observer agreement of presence of SMIC using high definition imaging and chromoendoscopy | Three years
Compare the difference between live endoscopic assessment and use of carefully selected endoscopic images to predict SMIC | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] Sidhu M, Shahidi N, Vosko S, van Hattem WA, Tate DJ, Bourke MJ. Incremental benefit of dye-based chromoendoscopy to predict the risk of submucosal invasive cancer in large nonpedunculated colorectal polyps. Gastrointest Endosc. 2022 Mar;95(3):527-534.e2. doi: 10.1016/j.gie.2021.11.032. Epub 2021 Dec 5. PMID 34875258